CLINICAL TRIAL: NCT00623324
Title: A Phase II, Dose Ranging, Randomized, Double Blind, Placebo-controlled, Multi-center, Pilot Study to Assess the Safety, Tolerability, Efficacy and Pharmacokinetics of Aplindore in Patients With Early Stage Parkinson's Disease
Brief Title: The Effects of Aplindore on the Treatment of Signs and Symptoms of Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ligand Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Aplindore-201; Aplindore-201
Record Dates: First submitted 2008-02-14; First posted 2008-02-26 (Estimated); Last update posted 2011-10-03 (Estimated); Status verified 2011-09

CONDITIONS: Early Stage Parkinson's Disease
MeSH Terms: interventions — aplindore fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Aplindore titrated to safe and tolerable dose
  Interventions: Drug: Aplindore
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aplindore — Tablets .05 - 5 mg BID dosing for 14 days
  Arms: 1
Drug: Placebo — Placebo tablets to match the number of active tablets
  Arms: 2

SUMMARY:
The purpose of this study is to demonstrate the safety, tolerability, efficacy and pharmacokinetics of aplindore in patients with early stage Parkinson's Disease (PD) who are not currently taking any dopamine agonists or who are able to wash off dopamine agonists for 14 days prior to baseline. Efficacy will be assessed using the UPDRS questionnaire including part 3 of the UPDRS (Motor). their level of sleepiness on a standardized rating scale (Epworth Sleepiness Scale) and their level of nausea daily.

Safety endpoints will include adverse events (AEs), clinical laboratory data, vital signs (blood pressure, orthostatic blood pressure and heart rate), ECGs, physical examinations and self rated scales.

DETAILED DESCRIPTION:
The purpose of this study is to demonstrate the safety, tolerability, efficacy and pharmacokinetics of aplindore in 5 groups of 8 patients each with early stage Parkinson's Disease (PD) based on Modified Hoehn and Yahr 1-3, who are not currently taking any dopamine agonists or who are able to wash off dopamine agonists for 14 days prior to baseline. Of the 8 patients in each cohort, 6 will be randomized to receive aplindore and two will receive placebo. The initial cohort of patients will be in the study unit from day -1 through day 15 (~2 weeks). After a review of safety labs and ECGs for Day -1, patients will begin twice a day dosing of investigational product on Day 1 with dosing to be given at within 30 minutes of completing breakfast and dinner, approximately 0700 and 1900.

A full UPDRS evaluation will be conducted at screen and on days -1, 7 and 14. In addition part 3 of the UPDRS (Motor) will be collected daily 2 hours after the morning dose of aplindore/placebo. At screening through discharge patients will be asked to self rate their level of sleepiness on a standardized rating scale (Epworth Sleepiness Scale) and their level of nausea daily 2 hours after the time of the morning dose of aplindore/placebo.

Safety endpoints will include adverse events (AEs), clinical laboratory data, vital signs (blood pressure, orthostatic blood pressure and heart rate), ECGs, physical examinations and self rated scales.

This study is a Phase II, dose-ranging, multi-center, placebo-controlled, double-blind, titration study to determine the safety, tolerability, efficacy and pharmacokinetics of aplindore in 5 groups of 8 patients each with early stage Parkinson's Disease (PD) based on Modified Hoehn and Yahr 1-3, who are not currently taking any dopamine agonists or who are able to wash off dopamine agonists for 14 days prior to baseline. Of the 8 patients in each cohort, 6 will be randomized to receive aplindore and two will receive placebo. The minimum number of patients required to initiate a cohort is 6 patients (4 randomized to aplindore and 2 to placebo). The patients in each cohort will be randomized in blocks of 4. Each site will recruit a full cohort of 6-8 patients per dose-titration regimen. There will be no sharing of cohorts/dose regimens across sites.

Early PD patients will be screened and 6-8 eligible patients will be housed in the study unit from day -1 through day 15 or until dismissed by the investigator. After a repeat of safety labs and ECG, patients will begin q12h dosing of investigational product (IP) with dosing to be given at within 30 minutes of completing breakfast and dinner, approximately 0700 and 1900 starting on Day 1. Doses will be escalated according to a predefined schedule. Two hours after each morning dose, a UPDRS part III will be performed. Safety will be ascertained by adverse events, ECGs, orthostatic vitals, physical and neurological exams, safety labs, Epworth Sleepiness Scale and Non Motor Symptoms Questionnaires. One blood sample for PK will be taken on each escalation day, 11 samples at steady state. ECGs and vital signs (semi-reclined and standing) will be collected each day at 2 hours post morning dosing. Adverse events will be collected throughout the inpatient stay. Patients will be down titrated upon reaching an intolerable dose. Patients on prior dopaminergic medications will resume their prior therapies on Day 15. Those patients not on prior dopaminergic medications will be down titrated over 5-7 days in the research clinic. Outpatient safety follow up will be 7-21 days after the last dose of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 30 years and above
* Must carry a diagnosis of idiopathic Parkinson's disease (PD), without any other known or suspected cause of parkinsonism, according to the UK Parkinson's Disease Society Brain Bank Clinical Diagnostic Criteria
* For early stage patients the initial diagnosis of PD must have been made within the 5 years prior to Screening with at least two or more of the following cardinal signs being present: bradykinesia, resting tremor, rigidity, and postural instability. In addition, they must not have developed motor complications from L-dopa use
* Early stage patients must be modified Hoehn & Yahr Stage 1 to 3 (inclusive)
* Must have a screening UPDRS (Part III) motor score of at least 10 Patients may be receiving amantadine, anticholinergics, COMT inhibitors and/or MAO-B inhibitor provided the dose was stable for at least 4 weeks prior to screening; dopamine agonists and/or L-dopa/carbidopa are permitted at screening but must be discontinued at least 14 days before baseline
* Good general health as determined by a thorough medical history and physical examination (including vital signs), 12-lead ECG and clinical laboratory tests
* Patients have clinical laboratory values within normal reference range or must not be clinically significantly abnormal as judged by the Investigator and approved by the Sponsor
* Patients taking prescription drug therapy or OTC medication for chronic medical conditions must be on stable doses for at least two (2) weeks prior to participation in the study and off any investigational drug for at least 60 days
* Females of childbearing potential must be using an acceptable method of contraception, have a negative urine pregnancy test at screening, and a negative urine pregnancy test on admission. Acceptable methods of contraception are oral, intrauterine, implantable, injectable contraceptives, double barrier methods or condoms impregnated with spermicide. After screening, patients using oral contraceptive methods of contraception must agree to add an additional method until 30 days following the last dose of study medication. Women on oral contraceptives must have been using them for at least one month prior to screening
* Male patients with partners of childbearing potential must use adequate contraception for 3 months after the study
* Female patients who have been surgically sterilized or have had a partial oopherectomy (i.e., one ovary intact) are eligible if they have a negative pregnancy test at screening and admission Be able to read, understand, and provide written/dated informed consent before enrolling in the study, and must be willing to comply with all study procedures;
* Patients must be willing and able to be confined to the clinical research unit as required by the protocol
* Patients must refrain from strenuous physical activity beginning 24 hours prior to screening and through the duration of the study
* Smokers may be enrolled if they have stable smoking habits

Exclusion Criteria:

* A Mini Mental State Examination (MMSE) score < 26
* History or clinical features consistent with an atypical parkinsonian syndrome
* History of surgical intervention for PD
* History of L-dopa-induced motor or non-motor complication
* History of severe allergic or anaphylactic reactions to any drug
* Clinically significant abnormal baseline ECG; QTcF > 450 msec for males, > 470 msec for females
* Recent history of severe dizziness or fainting due to postural hypotension; orthostatic blood pressure decrease defined as a drop in systolic BP of ≥ 40 mmHg and or a drop in diastolic BP of ≥ 20 mmHg following 5 minutes supine and 2 minutes standing in conjunction with symptoms.
* Evidence of clinically significant unstable allergic (except for untreated, asymptomatic, seasonal allergies at time of dosing), hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric or neurological disease
* History of cancer within 5 years of screening; except basal and squamous cell skin cancers and carcinoma in situ of the cervix
* Any condition that may affect drug absorption
* History of allergies, or known sensitivity, hypersensitivity, or adverse reaction to any drug similar to aplindore
* Pregnant or lactating females
* Recent history or current evidence of drug abuse or alcoholism; or withdrawal
* Introduction or dose change of hormone replacement therapy within 3 months

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Evaluation of safety and tolerability data | 3 weeks

SECONDARY OUTCOMES:
Change in UPDRS Motor (Part III) score, UPDRS Activities of Daily Living (ADL; Part II), the Non-Motor Symptoms Questionnaire, and the Epworth Sleepiness Scale (ESS) and nausea Likert Scale. | 3 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Miami Research Associates, Miami, Florida, United States